CLINICAL TRIAL: NCT02762539
Title: Omega3 PUFA in Head Trauam
Acronym: SMOFbrain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Omega 3 head injury
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Control group in which patients will follow our local protocol for TBI management without SMOF-lipid infusion
- SMOF group (Experimental): SMOF-lipid group in which patients will receive 0.5 g/Kg SMOF lipid 10% emulsion (Lipid emulsion for intravenous nutrition containing; 6% soybean oil / 6% medium chain triglycerides / 5% olive oil / 3%fish oil) daily over 12 hours starting once admitted to ICU for 7 days.
  Interventions: Drug: omega-3 enriched SMOF lipid emusion

INTERVENTIONS:
Drug: omega-3 enriched SMOF lipid emusion
  Arms: SMOF group

SUMMARY:
Traumatic brain injury (TBI) is major health problem that stands as a significant cause of death and permanent disability. TBI is considered as global public health epidemic. On pathophysiologic basis, TBI is described as occurring in two phases, primary and secondary. Once a primary insult occurs like trauma or ischemia, the secondary injury begins though main four mechanisms; ischemia, brain edema, axonal injury and neuro-inflammation. Omega-3 PUFAs (Polyunsaturated fatty acids) are postulated to have neuroregenerative properties with the ability to impact all four main mechanisms of the secondary injury Patients will be allocated into one of two groups through a random table generation; Control group in which patients will follow our local protocol for TBI management without SMOF-lipid infusion. SMOF-lipid group in which patients will receive 0.5 g/Kg SMOF lipid 10% emulsion (Lipid emulsion for intravenous nutrition containing; 6% soybean oil / 6% medium chain triglycerides / 5% olive oil / 3%fish oil) daily over 12 hours starting once admitted to ICU for 7 days

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate head trauma

Exclusion Criteria:

* sensitivity to SMOF lipid severe head trauama

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Glasgow coma scale after 48 hour of infusion | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Manşūrah, Dkahleya, Egypt

IPD SHARING:
Plan to Share IPD: Yes